CLINICAL TRIAL: NCT00400881
Title: Comparison Between Two Methods of Spontaneous Breathing Trial (SBT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Juan B. Figueroa-Casas, Associate Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E06040
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Results first posted 2012-05-17 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilation; weaning; respiratory failure; spontaneous breathing trial
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous PAP (CPAP) (No Intervention): CPAP (continuous positive airway pressure). 5 cm H2O.
- Automatic tube compensation (ATC) (Experimental): ATC is a new mode of ventilation being compared with traditional one (CPAP). ATC is a mode of ventilation of the same device (mechanical ventilator), not a new device. The pressure in this modes varies according the mechanical parameters of the respiratory system that are automatically calculated by this mode. This is the intervention arm.
  Interventions: Other: automatic tube compensation

INTERVENTIONS:
Other: automatic tube compensation — new mode of ventilation during spontaneous breathing trial. It is a mode of the same device (mechanical ventilator) where the pressure applied by the ventilator varies according to calculations o fthe mechanical properties of the respiratory system automatically performed by the ventilator.
  Arms: Automatic tube compensation (ATC)

SUMMARY:
To compare a new mode of mechanical ventilation, Automatic Tube Compensation (ATC) with a traditional one, Continuous Positive Airway Pressure(CPAP), on its effectiveness for detecting patients no longer needing mechanical ventilation.

DETAILED DESCRIPTION:
The ultimate goal of this proposal is to find the best way to rapidly and safely discontinue mechanical ventilation in patients recovering from respiratory failure.

It is common practice in these patients to perform trials of "spontaneous" breathing while still connected to the ventilator in order to assess their readiness to breathe without assistance. To help with this assessment, new mechanical modes have been incorporated to modern ventilators. A recently developed mode, called Automatic Tube Compensation, is designed for this purpose ("spontaneous" breathing). Whether this method is superior to traditional ones has not been established and the investigators intend to address this question.

The investigators aim to:

1. compare Automatic Tube Compensation vs. our traditional mode (Continuous Positive Airway Pressure) during spontaneous breathing trials in their efficacy to identify patients ready be successfully removed from mechanical ventilation
2. study which physiologic variables better predict successful discontinuation of mechanical ventilation in these two modes.

The investigators plan to prospectively randomize patients on mechanical ventilation at the point of weaning evaluation, to undergo spontaneous breathing trials with our current ventilatory mode (Continuous Positive Airway Pressure) or the new mode (Automatic Tube Compensation). Based on predefined physiologic and clinical variables, clinicians will decide whether patients are ready to be removed from mechanical ventilation. The proportions of successful discontinuation (no need to reinstitute mechanical ventilation) and the duration of the weaning period in both groups will be compared. During the spontaneous breathing trials, respiratory variables will be measured and compared between patients with successful vs. non successful discontinuation in order to evaluate their predictive value for successful outcome.

Mechanical ventilation is being used increasingly given our growing population with advanced age and multiple co morbidities and the rising volume of aggressive medical procedures. It is well known to be associated with medical complications and high health care costs. Reducing the duration of unnecessary mechanical ventilation while minimizing the risk of premature removal of needed assistance is the final objective of this project. Approaching this goal will decrease the adverse effects of this treatment and the cost of critical care.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older
* on mechanical ventilation at Thomason Hospital Intensive Care Unit for more than 24 hours
* about to undergo SBT by the current institutional protocol for weaning assessment ordered by their treating physician
* availability of informed consent from patient or next of kin

Exclusion Criteria:

* patients for whom a decision has been made not to reinstitute ventilatory assistance under any circumstance
* pregnancy
* patients not considered for discontinuation of mechanical ventilation on the day of SBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan B Figueroa-Casas, MD, Principal Investigator — Assistant Professor, Texas Tech University HSC
Locations (1):
- University Medical Center Hospital, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CPAP (Continuous Positive Airway Pressure): CPAP (continuous positive airway pressure)(standard mode of ventilation, non-intervention control group)
- Automatic Tube Compensation (ATC): ATC mode of ventilation (intervention, not-standard mode)
Period: Overall Study
Arm/Group | CPAP (Continuous Positive Airway Pressure) | Automatic Tube Compensation (ATC)
Started | 62 | 60
Completed | 62 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP (Continuous Positive Airway Pressure) | Automatic Tube Compensation (ATC) | Total
Number analyzed (Participants) | 62 | 60 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 50 | 105
  >=65 years | 7 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (19) | 52 (20) | 51 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 37 | 42 | 79
Region of Enrollment [Number; unit: participants]
  United States | 62 | 60 | 122

OUTCOME MEASURES:

1. Primary Outcome: Duration of Weaning Time
Description: Weaning time was determined as number of days from the day of the first SBT(spontaneous breathing trial) to the day of extubation. All patients were followed until extubation.
Time Frame: days
Population: All patients completing the SBT were analysed except for two patients in each group that were excluded from analysis per protocol due to re-intubation due to upper airway obstruction.
Measure: Mean (Standard Deviation); unit: days
Groups:
- CPAP: Continuous Positive Airway Pressure
- ATC (ATComp): Automatic Tube Compensation
Arm/Group | CPAP | ATC (ATComp)
Number analyzed (Participants) | 60 | 58
days | 0.18 (0.5) | 0.05 (0.3)

2. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration in days from day of intubation to day of extubation.
Time Frame: days
Population: Analysis per protocol. All patients completing the SBT were analysed except for two patients in each group that were excluded from analysis per protocol due to re-intubation due to upper airway obstruction.
Measure: Mean (Standard Deviation); unit: days
Groups:
- ATC (AT Comp): Automatic Tube Compensation
Arm/Group | CPAP | ATC (AT Comp)
Number analyzed (Participants) | 60 | 58
days | 4.9 (3.4) | 5.1 (4.2)

ADVERSE EVENTS:
Arm/Group | CPAP (Continuous Positive Airway Pressure) | Automatic Tube Compensation (ATC)
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/60
Other Adverse Events (participants affected / at risk) | 0/62 | 0/60

LIMITATIONS AND CAVEATS:
General ICU population.

Two subjects in each group were randomized and data collected but were not included in analysis per protocol due to needing re-intubation for upper airway obstruction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No